CLINICAL TRIAL: NCT02448667
Title: Energy Supplements to Improve Exercise Tolerance in Metabolic Myopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Astrid Emilie Buch, BSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-4-2014-014
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Glycogen Storage Disease Type III
MeSH Terms: conditions — Glycogen Storage Disease Type III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAXE Kondi - a sugary soft-drink (Experimental): 100 ml FAXE Kondi (10 grams of carbohydrates per 100 ml) is ingested every ten minutes during exercise plus 400 ml before exercise start.
  Interventions: Dietary Supplement: FAXE Kondi
- FAXE Kondi Free - a sugarfree soft-drink (Placebo Comparator): 100 ml FAXE Kondi Free (0 grams of carbohydrates per 100 ml) is ingested every ten minutes during exercise plus 400 ml before exercise start.
  Interventions: Dietary Supplement: Faxe Kondi Free

INTERVENTIONS:
Dietary Supplement: FAXE Kondi — Sucrose and glucose containing softdrink
  Arms: FAXE Kondi - a sugary soft-drink
Dietary Supplement: Faxe Kondi Free — Diet softdrink with artificial sweeteners aspartame and acesulfame potassium. Both sweeteners are approved for use as food additives in the European Union and by the FDA. Aspartame metabolism is well understood and normal doses does not affect plasma concentrations of lipids, amino acids, glucose levels, key regulatory hormones or skeletal muscle metabolism. Acesulfame Potassium is not metabolized in humans and is excreted as the parent compound in urine. Since the two artificial sweeteners does not affect skeletal muscle metabolism or blood glucose levels, and both compounds have a well documented safety profiles, FAXE Kondi Free is considered to be an ideal placebo soft drink in this study.
  Arms: FAXE Kondi Free - a sugarfree soft-drink

SUMMARY:
Patients suffering from the metabolic myopathy Glycogen Storage Disease type IIIa (GSDIIIa) have a problem releasing sugar stored in cells that is needed for energy production. This causes several systemic impairments, but only recently have the exercise-related symptoms in the muscles been examined. A previous study showed signs that intravenous infusion of glucose relieves some of these symptoms. The purpose of this study is to investigate in a randomized and placebo-controlled fashion whether oral ingestion of sugar can alleviate muscular symptoms in patients with GSDIIIa.

DETAILED DESCRIPTION:
It has recently been documented how patients with GSDIIIa have a moderate to severely reduced exercise capacity, and that exercise induces muscle pain and cramps. These symptoms are caused by the inability to mobilize skeletal muscle glycogen and are most likely the consequence of a severe energy deficiency within muscles. The study changed the phenotype of GSDIIIa, to include exercise-induced symptoms, which is a typical presentation in other metabolic myopathies. It also documented that exercise capacity was significantly improved while exercise-induced muscular symptoms were relieved by an intravenous glucose infusion. Based on these findings, this study wishes to investigate if oral ingestion of sucrose has the same effects on work capacity on a larger number of patients, in a randomized, placebo-controlled, cross-over setup. Ingestion of sucrose has the potential to be an effective, cheap and easily accessible dietary treatment of muscular symptoms in GSDIIIa.

ELIGIBILITY:
Inclusion Criteria:

* Genetically and/or biochemically verified GSDIIIa.
* 18 years or older.

Exclusion Criteria:

* Clinically significant cardiac or pulmonary disease.
* Pregnancy or lactation.
* Severe mental disorders or participants that are in other ways unable to understand the purpose of the trials.
* Subjects where the investigator assess that it is not possible or very difficult to place an intravenous catheters.
* Other conditions of the joints or skeletal muscle such as arthritis or sprains. If the condition is expected to resolve before the study inclusion period is stopped, the subject may be included at a later time.
* Moderate to severe muscle weakness, where the participants are not expected to complete 10 minutes of cycle-ergometry exercise at 70 % of VO2peak.
* Verified diabetes.
* Participation in other clinical trials that may interfere with the results.
* Medications that may interfere with the results or increase the risk of bleeding.
* Blood-clotting or bleeding disorders.
* Blood donation one month or less prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04-17 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
maximal work capacity | After up to 1 hour of bicycling on the 2nd and 4th day.
  Area Under the Curve (AUC) = resistance times duration of workout

SECONDARY OUTCOMES:
Peak oxygen consumption | After up to 1 hour of cycling on the 2nd and 4th day.
  (VO2peak)
Peak workload | After up to 1 hour of cycling on the 2nd and 4th day.
  (Wpeak)
Peak respiratory exchange ratio | After up to 1 hour of cycling on the 2nd and 4th day.
  (RER)
p-lactate | measured at rest and max on day 1, and before first dose of soft drink, before exercise and every 10 minutes during exercise at day 2 and 4.
  Analysis of blood sample
Heart rate | Continously during the cycle test (max. 1 hour) on the 2nd and 4th day
  pulsemonitoring
Borg score | Measured periodically during the cycle test (max. 1 hour) on the 2nd and 4th day
  Rate of percieved exertion

OTHER OUTCOMES:
Respiratory exchange ratio, RER | measured continously during the exercise test day 2 and 4.
  VO2/VCO2
p-glucose | measured at rest and max on day 1, and before first dose of soft drink, before exercise and every 10 minutes during exercise at day 2 and 4.
  Analysis of blood sample
Pain | Assessed on days 3 and 5 of the trial
  Pain assessed on a visual analog scale (VAS) with a scale of 0 to 10 cm
Fatigue | Assessed on days 3 and 5 of the trial
  Fatigue Severity Score (FSS)
p-Creatine kinase | measured on day 1, 3 and 5.
  To asses muscle damage
p-myoglobin | measured on day 1, 3 and 5.
  To asses muscle damage
p-ammonia | measured at rest and max on day 1, and before exercise, at 10 minutes, 20 min of exercise and at max on day 2 and 4.
  Analysis of blood sample
p-insulin | measured at rest and max on day 1 and before exercise and every 10 minutes during exercise at day 2 and 4.
  analysis of blood sample
p-glucagon | measured at rest and max on day 1, and before exercise, at 10 minutes, 20 min of exercise and at max on day 2 and 4.
  analysis of blood sample
p-catecholamines | measured at rest and max on day 1, and before exercise, at 10 minutes, 20 min of exercise and at max on day 2 and 4.
  analysis of blood sample
Hypoglycemic episodes | 2 hour observation after each of the two exercise test.
  Clinical observation as well as blood glucose levels monitored during exercise tests

CONTACTS AND LOCATIONS:
Overall Officials: Astrid E Buch, BSc Medicine, Principal Investigator — Copenhagen Neuromuscular Center
Locations (1):
- Copenhagen Neuromuscular Center, department 3342, Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kishnani PS, Austin SL, Arn P, Bali DS, Boney A, Case LE, Chung WK, Desai DM, El-Gharbawy A, Haller R, Smit GP, Smith AD, Hobson-Webb LD, Wechsler SB, Weinstein DA, Watson MS; ACMG. Glycogen storage disease type III diagnosis and management guidelines. Genet Med. 2010 Jul;12(7):446-63. doi: 10.1097/GIM.0b013e3181e655b6. PMID 20631546
- [Background] Van Hoof F, Hers HG. The subgroups of type 3 glycogenosis. Eur J Biochem. 1967 Oct;2(3):265-70. doi: 10.1111/j.1432-1033.1967.tb00134.x. No abstract available. PMID 5235982
- [Background] Coleman RA, Winter HS, Wolf B, Gilchrist JM, Chen YT. Glycogen storage disease type III (glycogen debranching enzyme deficiency): correlation of biochemical defects with myopathy and cardiomyopathy. Ann Intern Med. 1992 Jun 1;116(11):896-900. doi: 10.7326/0003-4819-116-11-896. PMID 1580445
- [Background] Preisler N, Pradel A, Husu E, Madsen KL, Becquemin MH, Mollet A, Labrune P, Petit F, Hogrel JY, Jardel C, Maillot F, Vissing J, Laforet P. Exercise intolerance in Glycogen Storage Disease Type III: weakness or energy deficiency? Mol Genet Metab. 2013 May;109(1):14-20. doi: 10.1016/j.ymgme.2013.02.008. Epub 2013 Feb 19. PMID 23507172
- [Background] Haller RG, Vissing J. Spontaneous "second wind" and glucose-induced second "second wind" in McArdle disease: oxidative mechanisms. Arch Neurol. 2002 Sep;59(9):1395-402. doi: 10.1001/archneur.59.9.1395. PMID 12223025
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Preisler N, Laforet P, Madsen KL, Hansen RS, Lukacs Z, Orngreen MC, Lacour A, Vissing J. Fat and carbohydrate metabolism during exercise in late-onset Pompe disease. Mol Genet Metab. 2012 Nov;107(3):462-8. doi: 10.1016/j.ymgme.2012.08.019. Epub 2012 Aug 31. PMID 22981821
- [Background] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Background] Coyle EF. Carbohydrate supplementation during exercise. J Nutr. 1992 Mar;122(3 Suppl):788-95. doi: 10.1093/jn/122.suppl_3.788. PMID 1542049
- [Background] Maki DG, Kluger DM, Crnich CJ. The risk of bloodstream infection in adults with different intravascular devices: a systematic review of 200 published prospective studies. Mayo Clin Proc. 2006 Sep;81(9):1159-71. doi: 10.4065/81.9.1159. PMID 16970212
- [Background] Chattopadhyay S, Raychaudhuri U, Chakraborty R. Artificial sweeteners - a review. J Food Sci Technol. 2014 Apr;51(4):611-21. doi: 10.1007/s13197-011-0571-1. Epub 2011 Oct 21. PMID 24741154
- [Background] Marinovich M, Galli CL, Bosetti C, Gallus S, La Vecchia C. Aspartame, low-calorie sweeteners and disease: regulatory safety and epidemiological issues. Food Chem Toxicol. 2013 Oct;60:109-15. doi: 10.1016/j.fct.2013.07.040. Epub 2013 Jul 23. PMID 23891579
- [Background] Magnuson BA, Burdock GA, Doull J, Kroes RM, Marsh GM, Pariza MW, Spencer PS, Waddell WJ, Walker R, Williams GM. Aspartame: a safety evaluation based on current use levels, regulations, and toxicological and epidemiological studies. Crit Rev Toxicol. 2007;37(8):629-727. doi: 10.1080/10408440701516184. PMID 17828671
- [Background] EFSA ANS Panel (EFSA Panel on Food Additives and Nutrient Sources added to food), 2013. Scientific Opinion on the re-evaluation of aspartame (E 951) as a food additive. EFSA Journal 2013;11(12):3496, 263 pp. doi:10.2903/j.efsa.2013.3496
- [Background] Harris RA. Carbohydrate metabolism I: Major metabolic pathways and their control. In: Devlin TM, ed. Textbook of biochemistry with clinical correlations, 6th ed Wiley-Liss, 2006:581-635
- [Background] DiMauro S, Hays AP, Tsujino S. Metabolic Disorders Affecting Muscle. In: Engel AG, Franzini-Armstrong C, eds. Myology, 3rd ed McGraw-Hill, 2004:1535-1558
- See also: Scientific Committee on Food. Re-evaluation of acesulfame K with reference to the previous SCF opinion of 1991. — http://ec.europa.eu/food/fs/sc/scf/out52_en.pdf